CLINICAL TRIAL: NCT01575574
Title: Magnetic Resonance With Gadoxetic Acid for the Diagnosis of Hepatocellular Carcinoma in Patients With Liver Cirrhosis. Evaluation of Its Impact for the Non-invasive Diagnosis
Acronym: PRIGA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIGA; 2011-005909-79 (EudraCT Number)
Record Dates: First submitted 2012-03-27; First posted 2012-04-11 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GADOXETIC ACID (Other): Is a non comparative study. a magnetic resonance will be done using gadoxetic acid : 0.025mmol/Kg
  Interventions: Drug: GADOXETIC ACID

INTERVENTIONS:
Drug: GADOXETIC ACID — all patients will have a magnetic resonance with gadobutrol as reference for diagnosis; in participants an additional magnetic resonance will be done with the new contrast agent to verify if the diagnostic can be done.

SUMMARY:
This is a study to evaluate the primovist as a new contrast agent useful to diagnostic of hepatocellular carcinoma

DETAILED DESCRIPTION:
The investigators plan to define the imaging patterns of hepatocellular carcinoma in cirrhotic patients when studied with gadoxetic acid magnetic resonance imaging including the dynamic phase and the hepatobiliary phase at 10 and 20 minutes after contrast injection and to evaluate the usefulness of liver magnetic resonance imaging with gadoxetic acid in the differentiation between benign and malignant nodules in the cirrhotic liver. To determine the diagnosis and clinical significance of the infracentimetric additional nodules detected in the hepatobiliary phase

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* patient with diagnosis of liver cirrhosis Child Pugh A-B
* Patients without previous hepatocellular carcinoma in whom ultrasound detects a suspicious hepatic lesion; solitary solid and well-defined nodule between 10 and 20mm
* patients in whom diagnosis of hepatocellular carcinoma is a clinical need prior to treatment indication
* patient that agree to participate signing informed consent form

Exclusion Criteria:

* Patients with poor liver function who would have undergone transplantation even without hepatocellular carcinoma diagnosis (Child-Pugh C)
* patients with previous diagnosis of hepatocellular carcinoma
* patients with significant comorbidities that could prevent the optimum therapeutic decision in case of positive diagnosis of hepatocellular carcinoma
* patients with severe clotting alterations that contraindicate the fine-needle biopsy -Patients with chronic kidney disease or glomerular filtration rate < 30 ml/min
* patients with contraindications to perform magnetic resonance imaging (pacemaker, claustrophobia...)
* Known hypersensitivity to study drugs or excipients
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
hepatocellular carcinoma diagnosed | 1 month
  Proportion of hepatocellular carcinoma diagnosed using gadoxetic acid magnetic resonance imaging (accuracy for diagnosis)

SECONDARY OUTCOMES:
magnetic resonance imaging sensitivity | 9 months
  magnetic resonance imaging sensitivity - number of patients that need fine-needle biopsy to the diagnosis.
  the patients would be followed until the diagnosis would be stablished. Is expected that this would be before 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Ayuso, Prof, PhD MD, Principal Investigator — Hospital Clínic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Barcelona, Spain